CLINICAL TRIAL: NCT03503656
Title: Evaluation and Usability of "Compuflo®" in Epidural Anesthesia for Obstetric and Gynecological Areas
Brief Title: "Compuflo®" in Epidural Space Identification
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Alessandro Di Filippo, Dr, Azienda Ospedaliero-Universitaria Careggi
Other Study IDs: CompuFlo AOUCareggi
Record Dates: First submitted 2018-04-05; First posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Anesthesia, Epidural; Analgesia, Epidural
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- CompuFlo: All the consecutive patients undergoing to an epidural catheter placement in Gynecological and Obstetric setting
  Interventions: Device: epidural catheter placement

INTERVENTIONS:
Device: epidural catheter placement — insertion of an epidural catheter using Compuflo System

SUMMARY:
Recently a computerized injection pump has been programmed with its own mathematical algorithm to measure on a digital display the pressure trend in the form of a continuous curve and it has been connected to an acoustic device that emits a sound at increasing frequencies during the progress of the epidural needle (Compuflo®, Milestone Scientific, Livingston, NJ); it has therefore been made capable of controlling the pressure at the injection point and adjusting the infusion rate according to a predetermined maximum value using the registered Dynamic Pressure Sensing (DPS) technology.

The Compuflo® system guarantees feedback on simultaneous and continuous pressure data, both visual and auditory, identifying and differentiating the different types of tissue. This safe and effective feedback helps medical personnel to identify the epidural space with greater accuracy and alerts them if the needle moves into the identified position.

The aim of the study was to verify the efficacy and usability of the Compuflo® system in a clinical setting.

The setting was the area of gynecology and obstetrics at a tertiary referral level University Hospital.

All the consecutive patients undergoing to an epidural catheter placement with Compuflo® were collected until to a sample size of 140 patients.

Primary endpoint was the number and percentage of successes in the placement of epidural catheters with Compuflo® Epidural. Secondary endpoints were: the number and percentage of accidental dural punctures during epidural catheter placement; the number of attempts aimed at the correct positioning of the epidural catheter; the measurement of procedure time duration; the measurement of pressure in the interspinous ligament, in the yellow ligament and within the epidural space; the measurement of volume of saline injected by Compuflo® to identify the epidural space.

ELIGIBILITY:
Inclusion Criteria:

signed informed consent to procedure more than 18 years of age

Exclusion Criteria:

NO

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the consecutive patients in gynecological and obstetric setting of a tertiary referral University Hospital submitted to epidural catheter insertion with CompuFlo® System
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
was the number of successes | 18 months
  number

SECONDARY OUTCOMES:
the number of accidental dural punctures | 18 months
  number
the number of attempts | 18 months
  number
procedure time duration | 18 months
  seconds
measurement of pressure in the interspinous ligament, in the yellow ligament and within the epidural space | 18 months
  mmHg
measurement of volume of saline injected by Compuflo® | 18 months
  ml

REFERENCES:
- [Background] Choi PT, Galinski SE, Takeuchi L, Lucas S, Tamayo C, Jadad AR. PDPH is a common complication of neuraxial blockade in parturients: a meta-analysis of obstetrical studies. Can J Anaesth. 2003 May;50(5):460-9. doi: 10.1007/BF03021057. PMID 12734154
- [Background] Lechner TJ, van Wijk MG, Maas AJ, van Dorsten FR, Drost RA, Langenberg CJ, Teunissen LJ, Cornelissen PH, van Niekerk J. Clinical results with the acoustic puncture assist device, a new acoustic device to identify the epidural space. Anesth Analg. 2003 Apr;96(4):1183-1187. doi: 10.1213/01.ANE.0000052382.04446.42. PMID 12651681
- [Background] Ghelber O, Gebhard RE, Vora S, Hagberg CA, Szmuk P. Identification of the epidural space using pressure measurement with the compuflo injection pump--a pilot study. Reg Anesth Pain Med. 2008 Jul-Aug;33(4):346-52. doi: 10.1016/j.rapm.2008.01.012. PMID 18675746